CLINICAL TRIAL: NCT04782921
Title: Clinical Outcomes of Papillae Tunneling Techniques in the Treatment of Isolated Intrabony Defects - a Prospective, Double Blind, Randomised Clinical Trial
Brief Title: Papillae Tunneling Techniques in the Treatment of Isolated Intrabony Defects
Acronym: PTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKCLjubljana
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis Complex; Xenograft Model

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel 40 (Experimental): Application of Gel 40
  Interventions: Device: Xenogenic bone graft material
- Gen-Os (Active Comparator): Application of Gen-Os
  Interventions: Device: Xenogenic bone graft material

INTERVENTIONS:
Device: Xenogenic bone graft material — After access to the periodontal defect via straight incision in vestibulum, at the mucogingival border or short releasing incision on adjacent tooth, Gel 40 (a mixture of collagen gel and xenogenic bone particles) or Gen-Os (pure xenogenic bone particles) will be inserted.

SUMMARY:
Papillae tunneling techniques (PTT) are a new approach toward regeneration of isolated intrabony defects. Compared to regular papillae preservation techniques, PTT rely on complete preservation of involved interdental papillae, providing optimal healing environment for periodontal wound. Surgical access is therefore gained either by vertical incision in vestibulum, or by short releasing incision on adjacent tooth. Interdental tissue is then carefully raised in a full thickness manner by tunneling instruments, root surface thoroughly cleaned by the ultrasound scaler or Gracey curettes and defect filled with the biomaterial of choice.

While the success and aesthetic results of non-incised papillae techniques are well documented, no paper so far compared clinical results of papillae preservation techniques with different biomaterials.

Therefore, the aim of our study is to compare gain of clinical attachment level (defined by sum of pocket probing depth and recession) to regular papillae preservation techniques, and to prove non-inferiority of Gel 40® (collagen matrix, loaded with micronized heterologous bone) to Gen-Os® (granulated cortico-cancellous heterologous bone mix).

Secondary objectives include analysis of aesthetic parameters - differences in recession and tip of the papillae location before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis stage III/IV
* at least one periodontal lesion with pocket probing depth > 5 mm, limited by 2 or more bone walls and intrabony component > 3 mm.
* good oral hygiene with plaque index and sulcular bleeding index < 30%.
* systemically healthy
* smokers and non-smokers

Exclusion Criteria:

* systemic diseases that contraindicate the treatment,
* on medications that affects periodontal healing
* pregnant or lactating women
* one wall intrabony defects
* defects that involve buccal and lingual side of the tooth
* tooth with incorrect endodontic treatment or restoration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change (CALC) | 6 and 12 months
  To evaluate the clinical attachment level change (CALG) in reconstructive periodontal treatment of isolated intrabony defects, using papillae preservation techniques and different biomaterials (Gel 40®, Gen-Os®).

SECONDARY OUTCOMES:
Wound closure (WC) | 1 week
  To determine if the early wound healing is dependent on the treatment choice.
Tip of papillae | 6 and 12 months
  To determine aesthetic result by measuring papillae tip position

OTHER OUTCOMES:
Probing pocket depth (PPD) | 6 and 12 months
  Measured with periodontal probe

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Faculty of Medicine, Ljubljana
  - University Dental Clinic, Ljubljana

REFERENCES:
- [Derived] Kobe T, Povsic K, Gaspersic R. Prehydrated collagenated cortico-cancellous heterologous bone gel and papillae tunneling for isolated intrabony defects: 12-month noninferiority trial. Clin Exp Dent Res. 2024 Feb;10(1):e853. doi: 10.1002/cre2.853. PMID 38345463